CLINICAL TRIAL: NCT07374653
Title: Online Cognitive Behavioural Therapy for Adolescents With Depression - A Randomized Controlled Trial
Brief Title: Online Self-healing Program
Acronym: iCBT-A
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HU-STA-00001939
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Mild to Moderate Depressive Symptoms

STUDY DESIGN:
Intervention Model Description: A clustered randomized controlled two-arm parallel-group trial will be adopted. Eligible adolescents will be openly recruited into activity groups from collaborating secondary schools. The activity groups are randomly allocated to the intervention groups and a control group on 1:1 ratio. Intervention group will receive iCBT-A. While the control group will receive online relaxation program (i.e., iRelaxation). Participants will complete the same online assessment tools at pre-intervention, post-intervention, and 3-month follow-up periods.
  Participants will receive weekly text and voice messages from student counsellors to promote adherence. In case, participants need more intensive support and individual counselling, participants, after giving their consent, will be referred by student counsellors to school social work services or counselling service of local social service by student counsellors. All student counsellors will be supervised by an experienced social worker and/or counsel
Who Masked: Investigator
Masking Description: A research staff, who does not involve in the group allocation and delivery of group interventions, conduct the intervention outcomes assessment of the participants before and after the intervention and 3-months follow-up. Actually, participants will complete the same online assessment tools at pre-intervention, post-intervention, and 3-month follow-up periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online cognitive behavioural therapy (Experimental): The online cognitive behavioural therapy (iCBT-A) offers six self-learning modules that participants can access via computer or smartphone to learn various CBT skills for managing emotional distress.
  Interventions: Behavioral: Online Cognitive Behaviural Therapy
- Online relaxation (Active Comparator): The online relaxation programme (iRelaxation) offers six self-learning modules that allow participants to use a computer or smartphone to learn various relaxation skills for managing emotional distress.
  Interventions: Behavioral: Online Relaxation

INTERVENTIONS:
Behavioral: Online Cognitive Behaviural Therapy — The online cognitive behavioural therapy (iCBT-A) provides six self-learning online modules for participants to learn via computer and/or smartphone a variety of CBT skills to manage their emotional distress. Participants in the intervention group will receive iCBT-A over a six-week period, completing one module per week. The iCBT-A includes the following topics: psychoeducation and normalization of the experience of mental health problems, and abdominal breathing (session 1); introduction to the basic concepts of CBT, identifying cognitive distortions and learning further relaxation techniques, including listening to relaxation music and imagery relaxation (sessions 2-3); learning cognitive restructuring skills (sessions 4-5); and developing a healthy lifestyle (session 6). Participants will receive weekly text and voice messages from student counsellors
  Arms: Online cognitive behavioural therapy
Behavioral: Online Relaxation — The online relaxation program (iRelaxation) provides six self-learning modules for participants to learn via computer and/or smartphone a variety of relaxation skills (such as breathing relaxation) to manage their emotional distress. Control group participants will receive the online relaxation program over a six-week intervention period, completing one module per week. The iRelaxation includes the following topics: abdominal breathing (sessions 1-2); imagery relaxation (sessions 3-4); and listening to relaxation music (sessions 5-6). Participants will receive weekly text and voice messages from student counsellors.
  Arms: Online relaxation

SUMMARY:
Background. Almost two thirds of adolescents experience a mental disorder before the age of 25. Among mental disorders, depression is one of the most common among young people aged between 15 to 24, with a prevalence of 13.5% to 15.8% worldwide and 13.2% in Hong Kong, which is alarming.

Cognitive behavioural therapy and online cognitive behavioural therapy has been shown to be effective on reducing depression. Also, online cognitive behavioural therapy has also been shown to be useful for people with mild to moderate depression. However, there is a lack of an effective short-term online cognitive behavioural therapy for adolescents with depression, named online cognitive behavioural therapy in Hong Kong.

Objectives: This study aims to explore the efficacy and effectiveness of a short-term online cognitive behavioural therapy for adolescents with depressive symptoms.

Hypothesis:

i. The online cognitive behavioural therapy, as compared to an online relaxation program, is significantly more effective on improving mental health, including reducing anxiety and depressive symptoms, and increasing psychological well-being for participants.

iii. The treatment outcomes, as stated in (i), are predicted by individual's uptake, adherence and dropout rate of online cognitive behavioural therapy.

Research Design. A multicentre blinded randomized controlled two-arm parallel-group trial will be adopted. Participating adolescents will be recruited from collaborating secondary schools. Using block randomization, subjects will be assigned in a 1:1 ratio to an online cognitive behavioural therapy and an online relaxation program. Both online cognitive behavioural therapy and online relaxation program will provide six online modules for participants to learn through computer and/or smartphone. Participants will complete the same online assessment tools at pre-intervention, post-intervention, and 2-month follow-up periods.

Subjects Inclusion Criteria. Subjects inclusion criteria includes: (a) aged between 12 and 18 years old; (b) students of a local collaborating secondary school; (c) having mild to moderate depressive symptoms as assessed with a standardized assessment tool, i.e. Chinese Depression Anxiety Stress Scale (DASS-Y; Cao et al., 2023) with a DASS Depression score of between 7 and 13; and (d) provide parental consent. Those with severe depression or at risk of suicide are excluded from this study.

Significance: This study aims to make a significant contribution to the development of an online cognitive behavioural therapy for Chinese adolescents with depressive symptoms. In particular, the online cognitive behavioural therapy could be used in secondary schools to serve those students with mental health problems who are reluctant to seek help from traditional face-to-face counselling.

DETAILED DESCRIPTION:
Introduction Almost two thirds (62.5%) of adolescents experience a mental disorder before the age of 25. Among mental disorders, major depressive disorder is one of the most common among young people aged between 15 to 24, with a prevalence of 13.5% to 15.8% worldwide and 13.2% in Hong Kong, which is alarming. Depression has negative effects on adolescents' mental and physical health and school performance, including suicide, alcohol and drug abuse, smoking, binge eating, diabetes, asthma and poor school performance.

Research evidences have consistently supported the efficacy and effectiveness of cognitive behavioural therapy on reducing depression in the Western, Asian, and Chinese societies.

Online cognitive behavioural therapy has been developed in which cognitive behavioural therapy is delivered via the internet helping individual to reduce their mental health problems using various skills developed by CBT. Online cognitive behavioural therapy has been reported to overcome the aforementioned barriers of traditional face-to-face psychological treatment by providing participants with flexible learning opportunities to read and learn the techniques and skills of cognitive behavioural therapy via an online platform that is accessible anytime, anywhere, anonymously, short-term, and in a structured manner. Research reviews have shown that online cognitive behavioural therapy is effective in reducing depression in adolescents with a small to medium effect size and the treatment effect of online cognitive behavioural therapy is comparable to that of face-to-face CBT.

Research Gap Currently, there is a lack of an effective short-term online cognitive behavioural therapy for adolescents with depression in Hong Kong and Chinese societies.

Objectives. This research project aims to design and investigate the intervention effects, uptake rate, and adherence rate and of a short-term online cognitive behavioural therapy for adolescents, named iCBT-A, with depressive symptoms in Hong Kong. Additionally, the predicting impact of uptake and adherence rates on treatment effects will also be investigated.

Hypothesis. i. The iCBT-A is significantly more effective than an online relaxation program on reducing depressive symptoms, and increasing psychological well-being for participants.

ii. The treatment outcomes, as stated in (i), are predicted by individual's uptake, adherence and dropout rate of iCBT-A.

Research Design. A clustered randomized controlled two-arm parallel-group trial will be adopted. Eligible adolescents will be openly recruited into activity groups from collaborating secondary schools. The activity groups are randomly allocated to the intervention groups and a control group on 1:1 ratio. Intervention group will receive iCBT-A. While the control group will receive online relaxation program (i.e., iRelaxation). Participants will complete the same online assessment tools at pre-intervention, post-intervention, and 2-month follow-up periods.

Participants will receive weekly text and voice messages from student counsellors to provide support and promote adherence. In case, participants need more intensive support and individual counselling, participants, after giving their consent, will be referred by student counsellors to school social work services or counselling service of local social service by student counsellors. All student counsellors will be supervised by an experienced social worker and/or counsellor of this project.

Special measures are implemented to reduce social stigma among secondary school students. Specifically, if there are six classes in Form 3, there will be six activity groups. These six groups will be randomly assigned to either the intervention group or the control group. Thus, three groups will be in the intervention group, while the other three will be in the control group. To reduce social stigma within the same class, non-eligible students studying in the same class as eligible students will receive the same iCBT-A or iRelaxation. For example, if eligible students in F.3A are assigned to the intervention group, the entire class of F.3A, including both eligible and non-eligible students, will receive the same iCBT-A. However, only outcome data from eligible students will be included in the final analysis.

Subjects Inclusion Criteria.

1. aged between 12 and 18 years old;
2. students of a local collaborating secondary school and/or youth service units;
3. having mild to moderate depressive symptoms as assessed with a standardized assessment tool, i.e. Chinese Depression Anxiety Stress Scale (DASS-Y) with a DASS Depression score of between 7 and 13; and
4. provide parental consent.

Exclusion criteria:

Those with severe depression (i.e., a DASS Depression score 14 or more) or at risk of suicide are excluded from this study.

Sample Size Estimation. Sample size is calculated using G*Power 3.1.1 software. Recent studies on iCBT suggest a small to medium effect size in reducing depression and anxiety (Hedges' g between 0.21 and 0.51). This study aims to demonstrate a small to medium effect size (i.e. Hedges' g = 0.30) with a statistical power of 0.80. A minimum sample size of 140 participants is required. In this study, a dropout rate of 40% is considered, and 200 participants will be recruited.

Intervention Group. An iCBT-A provides six self-learning modules for participants to learn via computer and/or smartphone a variety of CBT skills to manage their emotional distress. Intervention group participants will receive iCBT-A within a 6-weeks intervention period. The iCBT-A includes the following topics: psychoeducation and normalization of the experience of mental health problems, and abdominal breathing (session 1); introduction to the basic concepts of CBT, identifying cognitive distortions and learning further relaxation techniques, including listening to relaxation music and imagery relaxation (sessions 2-3), learning cognitive restructuring skills (sessions 4-5), and developing a healthy lifestyle (session 6). Participants will receive weekly text and voice messages from student counsellors.

Control Group. The iRelaxation provides six self-learning modules for participants to learn via computer and/or smartphone a variety of relaxation skills (such as breathing relaxation) to manage their emotional distress. Control group participants will receive the online relaxation program within a 6-weeks intervention period, with one module be completed per week. The iRelaxation includes the following topics: abdominal breathing (sessions 1-2), imagery relaxation (sessions 3-4), and listening to relaxation music (sessions 5-6). Participants will receive weekly text and voice messages from student counsellors.

Outcome Assessment Tools. The primary intervention outcome is improvement in mental health, including depression, anxiety and stress, assessed with the 21-item DASS-Y which has been demonstrated good validity and reliability (α = 0.80 for anxiety subscale, 0.83 for depression subscale, 0.82 for stress subscale, and 0.92 for whole scale).

The secondary intervention outcome is improvement in psychological well-being and stress reduction, which are assessed by:

The Chinese Flourishing Scale (FS) is an 8-item self-reported scale to assess psychological well-being, which has been shown satisfactory validity and internal consistency (Cronbach's α = 0.88).

The Adolescent Self-Rating Life Events (ASLEC) is a 27-item self-reported scale to assess stress reduction, which has been shown satisfactory validity and internal consistency (Cronbach's α = 0.92).

The Chinese Hope Scale (HOPE) is a 12-item scale to assess participants' self-reported hope with good validity and reliability (Cronbach's α = 0.81).

Ethical Approval. The ethical considerations of this study were evaluated and approved by the Research Committee of City University of Hong Kong. Written informed consent was obtained from all participants and their parents on or before the day of the pre-treatment assessment.

Data Analysis. An analysis will be performed in accordance with the intent-to-treat principle using multiple imputation method analysis for any missing data. Between group intervention effects will be investigated by using repeated measures of linear mixed model for repeated measures. In the linear mixed model, time, group, and time × group interactions were entered as fixed effects, with a random intercept for the subject. Effect sizes (Hedges' g) are calculated, with values of 0.2, 0.5, and 0.8 considered as small, medium, and large respectively. The predictive values of individual adherence, dropout and uptake rates of iCBTs are analysed using multiple linear regression analysis, with improved outcome assessment scores as dependent variables.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 12 and 18 years old;
2. students of a local collaborating secondary school and/or youth service units;
3. having mild to moderate depressive symptoms as assessed with a standardized assessment tool, i.e. Chinese Depression Anxiety Stress Scale (DASS-Y; Cao et al., 2023) with a DASS Depression score of between 7 and 13; and
4. provide parental consent.

Exclusion Criteria:

Those with severe depression (i.e., a DASS Depression score 14 or more) or at risk of suicide are excluded from this study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Chinese Depression Anxiety Stress Scale (DASS-Y) | DASS-Y will be used before intervention, after 6 weeks intervention, and 2-month follow-up.
  The DASS-Y is a 21-item scale to assess participant's self-reported mental health problems including depressive symptoms, anxiety symptoms and stress, with good validity and reliability (α = 0.80 for anxiety subscale, 0.83 for depression subscale, 0.82 for stress subscale, and 0.92 for whole scale; Cao et al., 2023). Each item (e.g. I felt down-hearted and blue) is scored from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). The scores are summed over the items with higher scores indicating a higher severity of symptoms. Each DASS-Y subscale score ranges from 0 to 21, while the DASS-Y total score ranges from 0 to 63.

SECONDARY OUTCOMES:
Chinese Flourishing Scale (FS) | FS will be used before intervention, after 6 weeks intervention, and 2-month follow-up.
  The Chinese Flourishing Scale (FS) is an 8-item self-reported scale to assess psychological well-being, which has been shown satisfactory validity and internal consistency (Cronbach's α = 0.88; Tong & Wang, 2017). Each itme (e.g. (I lead a purposeful and meaningful life) is rated with a score on a 4-point scale which ranges from "1" (strongly disagree) to "7" (strongly agree). The FS total scores range from 8 to 56, with higher scores indicating greater meaning and fulfillment.
Adolescent Self-Rating Life Events (ASLEC) | ASLEC will be used before intervention, after 6 weeks intervention, and 2-month follow-up.
  The Adolescent Self-Rating Life Events (ASLEC) is a 27-item self-reported scale to assess stress reduction, which has been shown satisfactory validity and internal consistency (Cronbach's α = 0.92; Liu et al., 1997). It covers 6 domains (interpersonal, academic, punishment, loss, health, other). Each item (e.g. Failure in an exam) is rated on a 6-point scale. The impact intensity of each item is rated using a five-point scale, ranging from '1 = no impact' to '5 = extremely severe'. If an event does not occur, it is rated as '0'.
Chinese Hope Scale (HOPE) | Chinese Hope Scale (HOPE) will be used before intervention, after 6 weeks intervention, and 2-month follow-up.
  The Chinese Hope Scale (HOPE) is a 12-item scale to assess participants' self-reported hope in two dimensions, i.e., agency (i.e., goal-directed energy) and pathways (i.e., planning to accomplish goals) with good validity and reliability (Cronbach's α = 0.81; 0.70 and 0.76 for the Hope total scale, agency subscale and pathway subscale; Ho et al., 2010). Each item (e.g. I can think of many ways to get out of a jam) is answered using an 4-point scale ranging from "1" (definitely false) to "4" (definitely true). The scores are summed over the items, ranging from 12 to 48. A higher score indicates a higher level of hope.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangwei Wanli School, Shenzhen, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Naudet C, Bystricky J, Carroll J, Gordon J, Hallman T, Igo G, Kirk P, Krebs GF, Lallier E, Landaud G, Letessier-Selvon A, Madansky L, Matis HS, Miller D, Roche G, Schroeder L, Seidl PA, Wang ZF, Welsh R, Yegneswaran A. Threshold behavior of electron pair production in p-Be collisions. Phys Rev Lett. 1989 Jun 5;62(23):2652-2655. doi: 10.1103/PhysRevLett.62.2652. No abstract available. PMID 10040053
- [Result] Bond MG, Workman G, Martland J, Clinkard JE, Carey BM, Rothwell RI, Joslin CA, Heron DA. Dosimetric considerations in the treatment of inoperable endometrial carcinoma by a high dose rate afterloading packing technique. Clin Oncol (R Coll Radiol). 1997;9(1):41-7. doi: 10.1016/s0936-6555(97)80060-x. PMID 9039813
- [Result] Toth JC. Is stress at hospital discharge after acute myocardial infarction greater in women than in men? Am J Crit Care. 1993 Jan;2(1):35-40. PMID 8353576
- [Result] Lui AS, Arnold JM. Response of large superficial dorsal hand veins to locally infused nitroglycerine in young, normal subjects. Can J Physiol Pharmacol. 1996 Sep;74(9):1034-8. PMID 8960395
- [Result] Hanin LG, Boucher KM. Identifiability of parameters in the Yakovlev-Polig model of carcinogenesis. Math Biosci. 1999 Aug;160(1):1-24. doi: 10.1016/s0025-5564(99)00029-2. PMID 10465929
- [Result] Atamas SP. Alternative splice variants of cytokines: making a list. Life Sci. 1997;61(12):1105-12. doi: 10.1016/s0024-3205(97)00243-9. PMID 9315502
- [Result] Petrides P. [Recommendations on the counseling of diabetics on the choice of career and occupational performance]. Dtsch Med Wochenschr. 1984 Sep 28;109(39):1499-501. No abstract available. German. PMID 6479049
- [Result] Perugia D, Basile A, Massoni C, Barletta V. Haemangiopericytoma in the distal third of the arm. Int Orthop. 1999;23(3):184-6. doi: 10.1007/s002640050343. PMID 10486035
- [Result] Aalto-Korte K, Turpeinen M. Pharmacokinetics of topical hydrocortisone at plasma level after applications once or twice daily in patients with widespread dermatitis. Br J Dermatol. 1995 Aug;133(2):259-63. doi: 10.1111/j.1365-2133.1995.tb02625.x. PMID 7547394
- [Result] Tong, K. K., & Wang, Y. Y. (2017). Validation of the Flourishing Scale and scale of positive and negative experience in a Chinese community sample. PloS one, 12(8), e0181616. https://doi.org/10.1371/journal.pone.0181616
- [Result] Liu, X., Liu, L., Yang, J., Chai, F., Wang, A., Sun, L., Zhao, G., & Ma, D. (1997). The Adolescent Self-Rating Life Events Checklist and its reliability and validity. Chinese Journal of Clinical Psychology, 5(1), 34-36
- See also: Related Info — https://doi.org/10.1371/journal.pone.0181616